CLINICAL TRIAL: NCT05141500
Title: SpO2 Accuracy of Noninvasive Pulse Oximeter Sensor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Sustainability Solutions (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CRD10302
Record Dates: First submitted 2021-11-23; First posted 2021-12-02 (Actual); Results first posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-11

CONDITIONS: Healthy; Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Intervention Model Description: Participants will be in a reclined position for the study. Reference sensors will be placed on each participant to evaluate the SpO2 accuracy and performance. Sensors may be placed on non-adjacent fingers to prevent optical crosstalk. Simultaneous data collection will be set up for devices under test. The data from the test devices will be collected by the sponsor or trained UCSF staff. Data will be collected for 1-2 second intervals data analysis. The SpO2 accuracy of the test devices will be evaluated over the oxygen saturation range between 70-100%.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Healthy adult participants (Experimental): All participants are enrolled in the test group and receive the noninvasive adhesive reprocessed pulse oximeter sensors
  Interventions: Device: STRYKER SUSTAINABILITY SOLUTIONS PULSE OXIMETERS

INTERVENTIONS:
Device: STRYKER SUSTAINABILITY SOLUTIONS PULSE OXIMETERS — Reprocessed noninvasive pulse oximeters
  * 1859 & 2329
  * MAX-A & MAX-N

SUMMARY:
The purpose of this clinical study is to validate the SpO2 accuracy of the Stryker Sustainability Solutions pulse oximetry sensors during non-motion conditions over the range of 70-100% SaO2 as compared to arterial blood samples assessed by CO-Oximetry. The end goal is to provide supporting documentation for the SpO2 accuracy validation of the reprocessed sensors.

DETAILED DESCRIPTION:
In this study, the level of oxygen within the blood will be reduced in a controlled manner by reducing the concentration of oxygen the participant breathes. The accuracy of a noninvasive pulse oximeter sensor will be assessed by comparison to the oxygen saturation measurements from a laboratory blood gas analyzer.

It is required that the Accuracy Root Mean Square (ARMS) performance of the Stryker pulse oximetry sensors will meet a specification of +/-3% or better in non-motion conditions for the range of 70 - 100% SaO2 (typically, saturation is determined once with air breathing and then at one of 6 levels, e.g. 94%, 90%, 85%, 80%, 75% and 70% saturation for about 30-60 seconds at each level), thereby demonstrating an acceptable SpO2 accuracy performance specification.

ELIGIBILITY:
Inclusion Criteria:

* Good general health with no evidence of pre-existing medical problems
* Fluent in both written and spoken English
* Must be able to review informed consent and is willing to comply with study procedures

Exclusion Criteria:

* Obesity (BMI >30)
* Known history of heart disease, lung disease, kidney or liver disease
* Prior diagnosis of asthma, sleep apnea, or use of CPAP
* Diabetes
* Clotting disorder
* Hemoglobinopathy or history of anemia that in the opinion of the investigators would make them unsuitable for study participation
* Any serious systemic illness
* Current smoker
* Any injury, deformity, or abnormality at the sensor sites that in the opinion of the investigator would interfere with the sensors working correctly
* History of fainting or vasovagal response
* History of sensitivity to local anesthesia
* Prior diagnosis of Raynaud's disease
* Unacceptable collateral circulation based on exam by investigators (Allen's test)
* Pregnant, lactating, or trying to get pregnant
* Unable or unwilling to provide informed consent, or unable or unwilling to comply with study procedures
* Any other condition which in the opinion of the investigators would make them unsuitable for the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip E Bickler, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Hypoxia Research Laboratory, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Data to be used by Sponsor only

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Adult Participants: All participants are enrolled in the test group and receive the noninvasive adhesive reprocessed pulse oximeter sensors
  STRYKER SUSTAINABILITY SOLUTIONS PULSE OXIMETERS: Reprocessed noninvasive pulse oximeters
  * Masimo pulse oximeter sensors, 1859 & 2329
  * Nellcor pulse oximeter sensors, MAX-A & MAX-N
Period: Overall Study
Arm/Group | Healthy Adult Participants
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Adult Participants
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 3
  Black or African American | 2
  Asian | 4
  Hispanic | 2
  Multiethnic | 1
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Sensor by Arms Calculation
Description: Percentage of SpO2 (oxygen saturation by pulse oximetry) measured by the Reprocessed Oximeter pulse oximetry sensors during non-motion conditions over the range of 70-100% SaO2 as compared to arterial blood samples assessed by CO-Oximetry. Accuracy root mean square (ARMS) between measured SpO2 and reference SaO2 (arterial oxygen saturation) must meet the 3% specification for each reprocessed pulse oximetry sensor style. Accuracy will be determined by comparing the noninvasive blood oxygen saturation measurement of the pulse oximeter to that obtained from a blood sample and calculating the arithmetic root mean square error (Arms) value. Standard deviation of the differences is computed as the precision. Square root of the sum of the squares of bias and precision is computed as the Arms Error value.
Time Frame: 1-2 hours
Measure: Number; unit: Root Mean Square Error (%)
Groups:
- Reprocessed MAX-N; Reprocessed MAX-A; Reprocessed 1859; Reprocessed 2329: All participants are enrolled in the test group and receive the noninvasive adhesive reprocessed pulse oximeter sensors.
Arm/Group | Reprocessed MAX-N | Reprocessed MAX-A | Reprocessed 1859 | Reprocessed 2329
Number analyzed (Participants) | 12 | 12 | 12 | 12
Root Mean Square Error (%) | 1.62 | 1.56 | 1.48 | 1.72

ADVERSE EVENTS:
Time Frame: 2 days
Arm/Group | Healthy Adult Participants
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/00/NCT05141500/Prot_SAP_001.pdf